CLINICAL TRIAL: NCT03937505
Title: A Phase 2 Multi-Center Safety and Efficacy Study of IS-001 Injection in Patients Undergoing Robotic Gynecological Surgery Using the da Vinci® Surgical System With Firefly® Fluorescent Imaging
Brief Title: A Safety and Efficacy Study of IS-001 Injection in Patients Undergoing Robotic Hysterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ISI-124804-2
Record Dates: First submitted 2019-04-29; First posted 2019-05-03 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Ureter Injury
Keywords: robotic-assisted surgery; minimally invasive surgery
MeSH Terms: interventions — IS 001

STUDY DESIGN:
Intervention Model Description: Stage A is a dose-cohort escalation to determine optimal efficacious dose, Stage B is an expanded safety and efficacy evaluation of the optimal dose with a no-drug safety control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose-escalation (Experimental): Dose-cohort escalation of single intravenous injection of IS-001 starting with 20 mg (n=8), escalating in 20 mg increments until optimal dose is determined.
  Interventions: Drug: IS-001
- Optimal dose-characterization (Experimental): Single intravenous injection of IS-001 at the optimal dose will be administered to subjects assigned to the treatment group. Safety control subjects will not receive any study drug but will undergo robotic surgery and all associated safety assessment clinical trial procedures.
  Interventions: Drug: IS-001; Drug: No treatment

INTERVENTIONS:
Drug: IS-001 — intravenous injection of IS-001 investigational drug
Drug: No treatment — no drug injection
  Arms: Optimal dose-characterization

SUMMARY:
This study evaluates the safety and efficacy of intravenous injection of IS-001 to aid in intraoperative ureter structure delineation. Stage A of the study will determine the safe optimal dose and Stage B will determine expanded safety and efficacy for intraoperative ureter structure delineation for the identified optimal dose in study participants.

DETAILED DESCRIPTION:
Injury to the ureter, the duct by which urine passes from the kidney into the bladder, is a well-known and serious complication of pelvic and abdominal surgery that frequently goes unrecognized intraoperatively. This study seeks to evaluate the safety and efficacy of intravenous IS-001 injection to improve surgeon ureter visualization during robotic-assisted surgery with the da Vinci® Surgical System and Firefly® imaging. Stage A will be a dose-escalation to determine the optimal dose for ureter visualization and Stage B will be an expanded safety and efficacy evaluation of the optimal dose. Stage B will include a no-drug safety control to evaluate the effects of surgery alone on the safety parameters of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Female subject is between the ages of 18 and 75, inclusive
2. Subject is scheduled to undergo robotic gynecological surgery using a da Vinci® surgical system with Firefly® fluorescent imaging
3. Subject is willing and able to provide informed consent
4. Subject is considered capable of complying with study procedures

Exclusion Criteria:

1. Subject is pregnant or nursing
2. Subject has known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection

4. Subject is already enrolled in another investigational study 5. Subject has any other condition or personal circumstance that, in the judgment of the Investigator, might interfere with the collection of complete quality data or represents an unacceptable safety profile

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Evaluate fluorescent intensity of ureter by signal to background analysis | 10 minutes
  Fluorescent intensity of ureter evaluated as signal to background
Evaluate fluorescent intensity of ureter by signal to background analysis | 30 minutes
  Fluorescent intensity of ureter evaluated as signal to background
Evaluate fluorescent intensity of ureter by signal to background analysis | 60 minutes
  Fluorescent intensity of ureter evaluated as signal to background

SECONDARY OUTCOMES:
Safety 12-Lead EKG Change from Baseline | 6 hours
  12-Lead EKG change from baseline in QTc
Incidence of abnormal blood work in tests results | 24 hours
  Safety hematology complete blood count laboratory assessments Change from Baseline
Incidence of abnormal blood work in tests results | 14 days
  Safety hematology complete blood count laboratory assessments Change from Baseline
Incidence of abnormal blood work in tests results | 24 hours
  Safety hematology comprehensive metabolic panel laboratory assessments Change from Baseline
Incidence of abnormal blood work in tests results | 14 days
  Safety hematology comprehensive metabolic panel laboratory assessments Change from Baseline
Incidence of abnormal urinalysis results | 14 days
  Routine urinalysis laboratory assessment change from baseline
Safety Adverse Events Monitoring | 14 days
  Drug related adverse events monitoring through 14-days
Pharmacokinetics Maximal Concentration (Cmax) of Drug Plasma Levels | 0, 1-2 hours and 2-3 hours
  Maximal concentration of investigational drug-plasma levels (Cmax)
Pharmacokinetics Area Under the Plasma Concentration Curve from Time Zero to Last Sampling (AUClast) | 0, 1-2 hours and 2-3 hours
  Area under the plasma curve from t(0) to last plasma sample
Pharmacokinetics Area Under the Plasma Concentration Curve from Time Zero Extrapolated to Infinity (AUCinf) | 0, 1-2 hours and 2-3 hours
  Area under the plasma curve from t(0) extrapolated to infinity
Pharmacokinetics Drug Plasma Clearance (CL) | 0, 1-2 hours and 2-3 hours
  Clearance of the investigational drug from plasma
Pharmacokinetics Terminal Elimination Half-life (t1/2) | 0, 1-2 hours and 2-3 hours
  Half-life of the investigational drug in plasma
Pharmacokinetics Apparent Volume of Distribution (Vz) | 0, 1-2 hours and 2-3 hours
  The apparent volume of distribution of the investigational drug
Ureter Identification Efficacy on a Nominal Scale | 10 minutes
  Independent reader assessment of ureter visibility of a 5 second video segment of the surgical field in both Firefly® and standard white light comparator mode on a nominal scale where 0=No and 1=Yes
Ureter Identification Efficacy on a Nominal Scale | 30 minutes
  Independent reader assessment of ureter visibility of a 5 second video segment of the surgical field in both Firefly® and standard white light comparator mode on a nominal scale where 0=No and 1=Yes
Ureter Identification Efficacy on a Nominal Scale | 60 minutes
  Independent reader assessment of ureter visibility of a 5 second video segment of the surgical field in both Firefly® and standard white light comparator mode on a nominal scale where 0=No and 1=Yes.
Ureter Delineation Efficacy as Length of Line Drawn in Millimeters | 10 minutes
  Independent reader assessment of ureter delineation on a still frame of the surgical field in both Firefly® and standard white light comparator mode. Length of line drawn on still frame where ureter is visible to independent reader is compared between imaging conditions.
Ureter Delineation Efficacy as Length of Line Drawn | 30 minutes
  Independent reader assessment of ureter delineation on a still frame of the surgical field in both Firefly® and standard white light comparator mode. Length of line drawn on still frame where ureter is visible to independent reader is compared between imaging conditions.
Ureter Delineation Efficacy as Length of Line Drawn | 60 minutes
  Independent reader assessment of ureter delineation on a still frame of the surgical field in both Firefly® and standard white light comparator mode. Length of line drawn on still frame where ureter is visible to independent reader is compared between imaging conditions.
Surgeon Confidence of Ureter Visibility Assessed Post-Dose by Three-point Likert-type Scale | 10 minutes post-dose
  Intra-operative surgeon rating of ureter visibility in surgical field in both Firefly® and standard white light comparator mode on a three point Likert-type scale where 0=No, 1=Uncertain and 2=Yes. Surgeon ureter visibility score will be compared between the two imaging conditions.
Surgeon Confidence of Ureter Visibility Assessed Post-Dose by Three-point Likert-type Scale | 30 minutes post-dose
  Intra-operative surgeon rating of ureter visibility in surgical field in both Firefly® and standard white light comparator mode on a three point Likert-type scale where 0=No, 1=Uncertain and 2=Yes. Surgeon ureter visibility score will be compared between the two imaging conditions.
Surgeon Confidence of Ureter Visibility Assessed Post-Dose by Three-point Likert-type Scale | 60 minutes post-dose
  Intra-operative surgeon rating of ureter visibility in surgical field in both Firefly® and standard white light comparator mode on a three point Likert-type scale where 0=No, 1=Uncertain and 2=Yes. Surgeon ureter visibility score will be compared between the two imaging conditions.
Surgeon Assessment of Relative Ureter Contrast Post-Dose on a Five-point Likert-type Scale | 10 minutes post-dose
  Intra-operative surgeon rating of relative ureter contrast in surgical field in Firefly® light mode on a five point Likert-type scale where 0=No Fluorescence, 1=Iso-Fluorescence, 2=Mild Fluorescence, 3= Moderate Fluorescence and 4=Strong Fluorescence. Surgeon contrast score will be compared to contrast scores at other time-points.
Surgeon Assessment of Relative Ureter Contrast Post-Dose on a Five-point Likert-type Scale | 30 minutes post-dose
  Intra-operative surgeon rating of relative ureter contrast in surgical field in Firefly® light mode on a five point Likert-type scale where 0=No Fluorescence, 1=Iso-Fluorescence, 2=Mild Fluorescence, 3= Moderate Fluorescence and 4=Strong Fluorescence. Surgeon contrast score will be compared to contrast scores at other time-points
Surgeon Assessment of Relative Ureter Contrast Post-Dose on a Five-point Likert-type Scale | 60 minutes post-dose
  Intra-operative surgeon rating of relative ureter contrast in surgical field in Firefly® light mode on a five point Likert-type scale where 0=No Fluorescence, 1=Iso-Fluorescence, 2=Mild Fluorescence, 3= Moderate Fluorescence and 4=Strong Fluorescence. Surgeon contrast score will be compared to contrast scores at other time-points.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Farnam, MD, Principal Investigator — Las Palmas Medical Center
Locations (3):
- United States (3):
  - George Washington University Hospital, Washington D.C., District of Columbia
  - St.David's Medical Center, Austin, Texas
  - Las Palmas Medical Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No